CLINICAL TRIAL: NCT03330197
Title: A Phase I/II Study of Ad-RTS-hIL-12, an Inducible Adenoviral Vector Engineered to Express hIL-12 in the Presence of the Activator Ligand Veledimex in Pediatric Brain Tumor Subjects
Brief Title: A Study of Ad-RTS-hIL-12 + Veledimex in Pediatric Subjects With Brain Tumors Including DIPG
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to slow accrual
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-103
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Brain Tumor; Diffuse Intrinsic Pontine Glioma
Keywords: DIPG; Glioblastoma; Anaplastic Astrocytoma; High Grade Glioma (HGG) Not Otherwise Specified (NOS); Supratentorial Tumor NOS
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioblastoma; Astrocytoma; Glioma | interventions — dipinacoline glutamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Closed (Experimental): Intratumoral Ad-RTS-hIL-12 freehand injection after tumor resection and oral veledimex (activator ligand) in pediatric patients with brain tumors.
  Interventions: Biological: Ad-RTS-hIL-12; Drug: Oral Veledimex - Arm 1 (Pediatric Brain Tumor)
- Arm 2 - Open (Experimental): Intratumoral Ad-RTS-hIL-12 stereotactic injection and oral veledimex (activator ligand) in pediatric patients with DIPG.
  Interventions: Biological: Ad-RTS-hIL-12; Drug: Oral Veledimex - Arm 2 (DIPG)

INTERVENTIONS:
Biological: Ad-RTS-hIL-12 — 2.0 x 10^11 viral particles (vp) per injection, one intratumoral injection of Ad-RTS-hIL-12
Drug: Oral Veledimex - Arm 1 (Pediatric Brain Tumor) — 1 dose level (10mg/day) 15 oral daily doses of veledimex
  Arms: Arm 1 - Closed
Drug: Oral Veledimex - Arm 2 (DIPG) — 2 dose levels (10mg/day, 20mg/day) 14 oral daily doses of veledimex
  Arms: Arm 2 - Open

SUMMARY:
This research study involves an investigational product: Ad-RTS-hIL-12 given with veledimex for production of human IL-12. IL-12 is a protein that can improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

The main purpose of this study is to evaluate the safety and tolerability of a single tumor injection of Ad-RTS-hIL-12 given with oral veledimex in the pediatric population.

DETAILED DESCRIPTION:
Eligible patients will be stratified to one of two arms, according to clinical indication for tumor resection. Pediatric patients who are scheduled for craniotomy and tumor resection will receive one dose of veledimex before the resection procedure. Ad-RTS-hIL-12 will be administered by free-hand injection. Patients will continue on oral veledimex for 14 days. This arm has been completed and is currently closed to enrollment.

Pediatric patients with diffuse intrinsic pontine glioma (DIPG) will receive Ad-RTS-hIL-12 by stereotactic injection and then will continue on oral veledimex for 14 days.

The study is divided into three periods: the screening period, the treatment period and the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≤ 21 years-of-age with the demonstrated ability to swallow capsules whole and who are willing to provide access to previously obtained biopsy results
2. Provision of written informed consent and assent, when applicable, for tumor resection, stereotactic surgery, tumor biopsy, sample collection, and/or treatment with study drug prior to undergoing any study-specific procedures
3. Arm 1: Evidence of recurrent or progressive supratentorial tumor, which has shown a > 25% increase in bi dimensional measurements by MRI or is refractory with significant neuro deterioration that is not otherwise explained with no known curative therapy, not in direct continuity with the ventricular system (e.g., there is physical separation between the tumor and ventricle, the tumor does not open directly into the ventricular system).

   Arm 2: Clinical presentation of DIPG and compatible MRI with approximately 2/3 of the pons included and without evidence of dissemination. Subjects should be ≥ 2 weeks and ≤ 10 weeks post standard focal radiotherapy (ie, dose of 5400 to 5960 cGy and maximum dexamethasone of 1 mg/m2/day)
4. At the time of registration, subjects must have recovered from the toxic effects of previous treatments, as determined by the treating physician.

   1. Targeted agents, including small-molecular tyrosine kinase inhibitors: 2 weeks
   2. Other cytotoxic agents: 3 weeks
   3. Nitrosoureas: 6 weeks
   4. Monoclonal antibody immunotherapies (eg, PD-1, CTLA-4): 6 weeks
   5. Vaccine-based and/or viral therapy: 3 months
5. On a stable or decreasing dose of dexamethasone for the previous 7 days
6. Able to undergo standard MRI scans with contrast agent before enrollment and after treatment
7. Have age-appropriate functional performance:

   1. Lansky score ≥ 40 or
   2. Karnofsky score > 50 or
   3. Eastern Cooperative Oncology Group (ECOG) score ≤ 2
8. Have adequate bone marrow reserves and liver and kidney function, as assessed by the following laboratory requirements:

   1. Hemoglobin ≥ 8 g/L
   2. Absolute lymphocyte count ≥ 500/mm3
   3. Absolute neutrophil count ≥ 1000/mm3
   4. Platelets ≥ 100,000/mm3 (untransfused [> 5 days] without growth factors)
   5. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for age
   6. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN for age
   7. Total bilirubin < 1.5 x ULN for age
   8. International normalized ratio (INR) and activated thromboplastin time within normal institutional limits
9. Male and female subjects of childbearing potential must agree to use a highly reliable method of birth control (expected failure rate < 1% per year) from the Screening visit through 28 days after the last dose of study drug. Women of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Radiotherapy treatment prior to the first veledimex dose:

   1. Focal radiation ≤ 4 weeks
   2. Whole-brain radiation ≤ 6 weeks
   3. Cranio-spinal radiation ≤ 12 weeks NOTE: Subjects in Arm 2 (ie, with DIPG) must be ≥ 2 weeks and ≤ 10 weeks after standard focal radiotherapy (dose of 5400 to 5960 cGy and maximum dexamethasone of 1 mg/m2/day)
2. Subjects with clinically significant increased intracranial pressure (eg, impending herniation or requirement for immediate palliative treatment) or uncontrolled seizures
3. Subjects whose body surface area (BSA) would expose them to < 75% or > 125% of the target dose
4. Known immunosuppressive disease, autoimmune condition, and/or chronic viral infection (eg, human immunodeficiency virus [HIV], hepatitis)
5. Use of systemic antibacterial, antifungal, or antiviral medications for the treatment of acute clinically significant infection within 2 weeks of first veledimex dose. Concomitant therapy for chronic infections is not allowed. Subjects must be afebrile prior to Ad-RTS-hIL-12 injection; only prophylactic antibiotic use is allowed perioperatively
6. Use of enzyme-inducing antiepileptic drugs (EIAEDs) within 7 days prior to the first dose of study drug
7. Other concurrent clinically active malignant disease, requiring treatment
8. Nursing or pregnant females
9. Prior exposure to veledimex
10. Use of medications that induce, inhibit, or are substrates of cytochrome p450 (CYP450) 3A4 within 7 days prior to veledimex
11. Use of heparin or acetylsalicylic acid (ASA). The use of systemic heparinization, or any ASA containing medications, is prohibited during active dosing with veledimex. Prophylactic heparin SC, per institutional protocol, or heparin when used for maintaining patency of an access port of a PICC line is permitted.
12. Presence of any contraindication for a neurosurgical procedure
13. Unstable or clinically significant concurrent medical condition that would jeopardize the safety of a subject and/or their compliance with the protocol

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (3):
- United States (3):
  - University of California San Francisco, Benioff Children's Hospital, San Francisco, California
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana- Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One Arm 2 subject was screened and enrolled but consent was withdrawn prior to Day 0.
Pre-assignment Details: All subjects in Arm 1 received 10mg daily of veledimex. A total of three subjects were assigned to Arm 2. One subject withdrew consent prior to any study procedures on Day 0 and received no treatment. A second subject was discontinued from the study due to a Serious Adverse Event (SAE) after the Ad-RTS-hIL-12 injection but prior to receiving veledimex. The third subject received veledimex at a dose of 5 mg/day, which was the body surface area (BSA)-adjusted dose.
Groups:
- Arm 1 - Closed: Intratumoral Ad-RTS-hIL-12 freehand injection after tumor resection and oral veledimex (activator ligand) in pediatric patients with brain tumors.
  Ad-RTS-hIL-12: 2.0 x 10^11 viral particles (vp) per injection, one intratumoral injection of Ad-RTS-hIL-12
  Oral Veledimex - Arm 1 (Pediatric Brain Tumor):
  * Planned: 1 dose level (10mg/day) 15 oral daily doses of veledimex
  * Actual: All patients received 1 dose level (10 mg/day veledimex)
- Arm 2 - Closed: Intratumoral Ad-RTS-hIL-12 stereotactic injection and oral veledimex (activator ligand) in pediatric patients with DIPG.
  Ad-RTS-hIL-12: 2.0 x 10^11 viral particles (vp) per injection, one intratumoral injection of Ad-RTS-hIL-12
  Oral Veledimex - Arm 2 (DIPG):
  * Planned:2 dose levels (10mg/day, 20mg/day)
  * Actual: 1 patient received 5 mg/day veledimex. The other patient did not receive veledimex due to SAE.
Period: Overall Study
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Started | 3 | 3
Treated With Ad-RTS-hIL-12 Injection | 3 | 2
Treated With Veledimex | 3 | 1
Did Not Receive Veledimex Treatment | 0 | 2
Received Veledimex Treatment | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline population includes every subject who received at least one dose of any study drug recorded in the Data Management (DM) database excluding screen failures. One patient in arm 2 withdrew consent prior to dosing and is considered a screen failure and one patient in Arm 2 only received Ad-RTS-hIL-12 (veledimex was not administered due to a serious adverse event.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Closed | Arm 2 - Closed | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Full Range); unit: years] | 16.1 [12.1 to 21.9] | 5.8 [5.7 to 5.9] | 12.1 [5.7 to 21.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
WHO High Grade at Baseline [Count of Participants; unit: Participants] — WHO grading of pediatric brain tumors range from Grade 1 (Low Grade) - Slow-growing, to Grade 4 (High Grade) - The most aggressive which grows and spreads rapidly and is difficult to treat. In this study all patients were high grade which means the tumor is already classified as aggressive and likely to spread and come back (recur) after treatment. These tumors have a poorer prognosis (outlook) than low-grade ones.
  Participants | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of Intratumoral Ad-RTS-hIL-12 and Veledimex as Measured by Dose Limiting Toxicities and Compliance.
Description: Dose Limiting Toxicities are defined as events that occur during the first 28 days (Day 0 - Day 28) that meets one of the following criteria:
  * Any local reaction that requires operative intervention and is felt to be attributable to study drug
  * Any local reaction that has life-threatening consequences requiring urgent intervention or results in death and is felt to be attributable to study drug
  * Any Grade 3 or higher non-hematologic adverse event that is at least possibly related to study drug and lasts ≥ 3 days
  * Nausea and vomiting will not be considered a DLT unless at least Grade 3 and refractory to antiemetics
  * Grade 3 or higher thrombocytopenia (< 50,000/mm3) at least possibly related to study drug
  * Any Grade 4 hematologic toxicity (except thrombocytopenia) that is at least possibly related to study drug and lasts ≥ 5 days
  * Transient neurological changes are expected in Arm 2 and will not be considered a DLT unless they last > 10 days
Time Frame: From Day 0 through Day 56
Population: The Full Analysis Set (FAS) or the OSP includes every subject who received at least one dose of any study drug recorded in the Data Management (DM) database excluding screen failures.
  • The data analysis for Adverse Events or other Safety variables will be performed on the OSP.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 2
Participants
  DLTs | 0 | 1
  AE leading to death | 0 | 0
  AEs leading to study discontinuation | 0 | 0
  AEs leading to study treatment discontinuation | 0 | 1
  AE leading to leading to study treatment dose reduction | 0 | 0
  Adverse events leading to study treatment dose interruption | 1 | 1
  Treatment emergent adverse events | 3 | 2

2. Secondary Outcome: To Measure the Veledimex in Blood and Brain Tumor by Using the LC-MS Method
Description: Veledimex brain concentration. Veledimex plasma concentration was below the limit of quantitation for most patients.
  Given the limited number of subjects enrolled and early closure of the study, complete assessment of veledimex in blood and brain tumor could not be determined.
Time Frame: From Day 0 through Day 15 of veledimex dosing
Population: Patients with available brain tumor results. Arm 2 patient result was below the level of quantitation (1.8 ng/mL). Arm 1 BLQ was 0.1 ng/mL. One patients was less than BLQ.
  Arm 2 patient plasma concentrations were not reported due to bioanalytical non-reproducibility. NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 1
ng/mL
  Brain tumor results (Day 0) | 0.172 [0.1 to 0.211] | NA [NA to NA] — For the one patient analyzed in Arm 2, the brain tumor concentration at Day 0 was Below the Quantitation Limit (BQL) of 1.80 ng/mL. All subsequent plasma concentrations for this patient were reported by the laboratory as Non-Reportable Results (NRR) and are therefore not available.
  Day 0 time of resection - veledimex plasma PK | 1.40 [1.00 to 1.86] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 1 predose- veledimex plasma PK | 1.02 [1 to 1.07] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 1 2 hr postdose- veledimex plasma PK | 11.64 [8.61 to 13.8] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 1 4 hr postdose- veledimex plasma PK | 5.66 [3.31 to 9.85] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 1 6 hr postdose- veledimex plasma PK | 5.64 [2.91 to 11.1] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 2 - veledimex plasma PK | 2.09 [1.4 to 2.92] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 14 predose- veledimex plasma PK | 4.39 [2.61 to 6.15] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 14 2 hr postdose - veledimex plasma PK | 36.83 [14.3 to 66.9] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 14 4 hr postdose - veledimex plasma PK | 19.80 [9.19 to 30.9] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 14 6 hr postdose - veledimex plasma PK | 7.63 [7.41 to 8.05] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.
  Day 15 24 hr postdose - veledimex plasma PK | 4.35 [3.13 to 5.03] | NA [NA to NA] — For the one patient who received veledimex and was analyzed, plasma concentration was reported by the lab as NRR (Non-Reportable Results). NRR (Non-Reportable Results) is the actual result reported from the central lab which was due to assay reagent expiration.

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from the first dose of the study drug to the date of death. Subjects were followed for up to 2 years.
Time Frame: 2 Years
Population: The Safety Population was defined as all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 2
participants
  Deceased | 2 | 1
  Alive | 0 | 1
  Unknown | 1 | 0

4. Secondary Outcome: Measure Immune Response of Ad-RTS-hIL-12 and Veledimex by a Quantitative Multiplex Immunoassay for Determination of IL-12 and IFNg Levels
Description: Samples for serum cytokine analysis were collected on Days 0, 3, 7, 14, and 28. For the results, participants who had samples analyzed were included in the "number analyzed" counts; however, values that were below the limit of quantitation (BLQ) were excluded from the calculation of mean and standard deviation.
Time Frame: Day 0, Day 3, Day 7, Day 14, and Day 28
Population: The Biomarker Evaluation Population (BEP) includes all subjects who received Ad-RTS-hIL-12 + at least one dose of their cohort-specific dose of veledimex who have adequate biomarker sample(s) at screening (baseline) and at least one non-missing follow-up biomarker assessment, excluding the disqualified assessments. All biomarker related data presentation will be based on the BEP unless specified otherwise. Note: In Arm 2, only 1 subject met this criteria.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 1
pg/mL
  Serum IFN-gamma - Day 0 | NA (NA) — All subjects had BLQ values at this time point. BLQ was reported as <2.4 pg/mL. | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <2.4 pg/mL.
  Serum IFN-gamma - Day 3: number analyzed (Participants) | 2 | 1
  Serum IFN-gamma - Day 3 | 4.4 (0) | 11.4 (0)
  Serum IFN-gamma - Day 7 | 6.4 (0) | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <2.4 pg/mL.
  Serum IFN-gamma - Day 14: number analyzed (Participants) | 2 | 1
  Serum IFN-gamma - Day 14 | NA (NA) — Two subjects had BLQ values at this time point. BLQ was reported as <2.4 pg/mL. | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <2.4 pg/mL.
  Serum IFN-gamma - Day 28: number analyzed (Participants) | 2 | 1
  Serum IFN-gamma - Day 28 | NA (NA) — Two subjects had BLQ values at this time point. BLQ was reported as <2.4 pg/mL. | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <2.4 pg/mL.
  Serum IL-12 - Day 0 | 12 (0) | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <1.6 pg/mL.
  1.6Serum IL-12 - Day 3: number analyzed (Participants) | 2 | 1
  1.6Serum IL-12 - Day 3 | 11.1 (2.1) | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <1.6 pg/mL.
  Serum IL-12 - Day 7 | 6.6 (4.7) | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <1.6 pg/mL.
  Serum IL-12 - Day 14: number analyzed (Participants) | 2 | 1
  Serum IL-12 - Day 14 | NA (NA) — Two subjects had BLQ values at this time point. BLQ was reported as <2.4 pg/mL. | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <1.6 pg/mL.
  Serum IL-12 - Day 28: number analyzed (Participants) | 2 | 1
  Serum IL-12 - Day 28 | 1.6 (0) | NA (NA) — Subject's result was BLQ at this time point. BLQ was reported as <1.6 pg/mL.

5. Secondary Outcome: Subjects With Ad-RTS-hIL-12 and Veledimex Related Adverse Events Will be Assessed for Safety by CTCAE v5.0
Description: Subjects with Ad-RTS-hIL-12 and veledimex related adverse events will be assessed for safety by CTCAE v5.0
Time Frame: 2 Years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 2
participants
  WHITE BLOOD CELL COUNT DECREASED (INVESTIGATIONS) | 2 | 2
  LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 2 | 2
  VOMITING (GASTROINTESTINAL DISORDERS) | 2 | 1
  HEADACHE (NERVOUS SYSTEM DISORDERS) | 2 | 1
  PYREXIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 2
  ANAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 2 | 0
  APHASIA (NERVOUS SYSTEM DISORDERS) | 1 | 1
  FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 | 1
  HYPONATRAEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 | 0
  NAUSEA (GASTROINTESTINAL DISORDERS) | 1 | 1
  PLATELET COUNT DECREASED (INVESTIGATIONS) | 2 | 0
  TACHYCARDIA (CARDIAC DISORDERS) | 0 | 2

6. Secondary Outcome: Best Overall Response by iRANO Criteria
Description: Best Overall Response was assessed using the immunotherapy Response Assessment for Neuro-Oncology (iRANO) criteria.
Time Frame: 2 Years
Population: The Efficacy Evaluable population is defined as all subjects who received at least 1 dose of study drug and had at least one post-treatment tumor assessment.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 3 | 2
participants
  Best Tumor Response SD | 0 | 2
  Best Tumor Response PD | 3 | 0
  Not Evaluable | 0 | 1

7. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) was defined as the time from the first documentation of a Complete Response (CR) or Partial Response (PR) to the first documentation of Progressive Disease (PD) or death due to any cause, whichever occurred first.
Time Frame: From the time of first response (CR or PR) until progression or death
Population: The analysis population for this measure included subjects from the Efficacy Evaluable population who achieved a Complete Response (CR) or Partial Response (PR).
Arm/Group | Arm 1 - Closed | Arm 2 - Closed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Arm 1: Intratumoral Ad-RTS-hIL-12 freehand injection after tumor resection and oral veledimex (activator ligand) in pediatric patients with brain tumors.
  Ad-RTS-hIL-12: 2.0 x 10^11 viral particles (vp) per injection, one intratumoral injection of Ad-RTS-hIL-12
  Oral Veledimex - Arm 1 (Pediatric Brain Tumor): 1 dose level (10mg/day) 15 oral daily doses of veledimex
- Arm 2: Intratumoral Ad-RTS-hIL-12 stereotactic injection and oral veledimex (activator ligand) in pediatric patients with DIPG.
  Ad-RTS-hIL-12: 2.0 x 10^11 viral particles (vp) per injection, one intratumoral injection of Ad-RTS-hIL-12
  Oral Veledimex - Arm 2 (DIPG): 2 dose levels (10mg/day, 20mg/day) 14 oral daily doses of veledimex
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=3) | Arm 2 (N=2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=3) | Arm 2 (N=2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (4) | 2 (5)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (3) | 2 (3)
ANAEMIA (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 2 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (2)
ALKALOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
ATAXIA (Nervous system disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
CANDIDA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FACIAL NERVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
FACIAL PARESIS (Nervous system disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1)
HEMIANOPIA (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPLEGIA (Nervous system disorders) | 0 (0) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (4)
MADAROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
OPTIC NERVE DISORDER (Eye disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 2 (2) | 0 (0)
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 0 (0) | 1 (1)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
VESSEL PUNCTURE SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (5)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the limited number of subjects enrolled and early closure of the study, complete assessment of safety and tolerability could not be determined. There was a wide range of adverse events reported and limited survival among the subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03330197/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03330197/SAP_001.pdf